CLINICAL TRIAL: NCT03938064
Title: Timing of Initiation of Luteal Phase Support in Poor Responders Undergoing IVF/ICSI: a Randomized Controlled Trial
Brief Title: Timing of Initiation of Luteal Phase Support in Poor Responders Undergoing IVF/ICSI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Collaborators: Ahmed Mahmoud Abdel-Rahim (Unknown)
Responsible Party: Principal Investigator, mostafa fouad gomaa, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Timing of initiation of luteal
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Infertility
Keywords: poor responders; IVF/ICSI; Luteal Phase Support; GnRH Antagonist Protocol
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Early start (Active Comparator): group will include 260 women with POR undergoing a trial of IVF/ICSI. This group will receive vaginal micronized progesterone pessaries from the day of ovum retrieval (OR).
  Interventions: Drug: Prontogest 400 mg vaginal pessaries
- Group Late start (Placebo Comparator): group will include 260 women with POR undergoing a trial of IVF/ICSI. This group will receive vaginal micronized progesterone pessaries 2 days after OR.
  Interventions: Drug: Prontogest 400 mg vaginal pessaries

INTERVENTIONS:
Drug: Prontogest 400 mg vaginal pessaries — natural progesterone in the form of vaginal suppositories 400 mg
  Other Names: placebo vaginal pessaries

SUMMARY:
It is already known that all stimulated IVF ICSI cycles needs luteal phase support for higher pregnancy rates The current study will focus on evaluating two different starting times of luteal phase support

DETAILED DESCRIPTION:
The optimal stimulation protocol for poor responder patients is a therapeutic challenge. However the lack of initial central down-regulation in early follicular phase and adequate prevention of premature luteinizing hormone (LH) surge in late follicular phase provide GnRH antagonist protocol as a potentially proper option for poor responders . Significant reduction in gonadotropin dosage and stimulation period could be achieved by antagonist protocol. Nevertheless, there are no significant differences in terms of clinical pregnancy and cancellation rates between the GnRH antagonist and agonist in poor responder patients .

a study evaluated the nonsupplemented luteal phase characteristics in patients undergoing ovarian stimulation with recombinant FSH and GnRH-antagonist cotreatment. With the administration of GnRH antagonist, luteolysis started prematurely because of excessive negative steroid feedback, resulting in suppressed pituitary LH release; low pregnancy rates were observed . In another study, the endometrium demonstrated abnormal development in oocyte donors who were stimulated with a GnRH-antagonist protocol but not supplemented in the luteal phase . Low luteal LH serum concentration and shortened luteal phase indicated the need for luteal phase supplementation in GnRH-antagonist IVF cycles .

Luteal phase support with hCG or progesterone after assisted reproduction results in an increased pregnancy rates . Natural micronized progesterone is not efficient if taken orally . The oral dydrogesterone (DG) might be sufficient for luteal supplementation in IVF cycles, however more large randomized controlled trials are needed before a conclusion about oral DG can be drawn . Vaginal and IM progesterone seem to have comparable implantation and clinical pregnancy rates and delivery rates . Concomitant use of E2 with progesterone after stimulation with rec-FSH and GnRH antagonist does not enhance the probability of pregnancy . Although there have been attempts to introduce GnRH agonist as a novel LPS in stimulated IVF cycles to improve PR, it is too early to adopt this approach across the board .

Timing of LPS remains the subject of debate, current clinical practice involves beginning LPS on different days. Starting progesterone on the day before oocyte retrieval or waiting until day 6 after retrieval may result in lower pregnancy rates. There appears to be a window for progesterone start time between the evening after oocyte retrieval and day 3 after oocyte retrieval. Although some have suggested a potential benefit in delaying vaginal progesterone starting time to 2 days after oocyte retrieval. It remains unclear whether pregnancy rates can be improved by delaying the progesterone initiation until the end of this progesterone window to avoid endometrial advancement . Additional randomized clinical trials are needed to better define progesterone start time for luteal support, particularly for vaginal progesterone, which may more rapidly advance the endometrium .

2. OBJECTIVES Research hypothesis: in poor responder women undergoing IVF/ICSI, starting luteal phase support (LPS) on day of ovum retrieval or 2 days later may have similar pregnancy rates.

Research question: in poor responder women undergoing IVF/ICSI does start of LPS on day of ovum retrieval or 2 days later lead to similar pregnancy rates? Aim of the study: to compare starting luteal phase support at day of ovum retrieval and 2 days after ovum retrieval in terms of ongoing pregnancy rates in POR patients undergoing IVF/ICSI cycles using GnRH antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

- At least two of the following three features must be present Advanced maternal age (40 years) or any other risk factor for Poor Ovarian Response

A previous POR (≤3 oocytes with a conventional stimulation protocol):

An abnormal ovarian reserve test (ORT): (i.e. AFC< 5-7 follicles or AMH 0.5-1.1ng/ml Two episodes of POR after maximal stimulation are sufficient to define a patient as poor responder in the absence of advanced maternal age or abnormal ORT By definition, the term POR refers to the ovarian response and, therefore, one stimulation cycle is considered essential for the diagnosis of POR, However, patients over 40 years of age with abnormal ORT may be classified as poor responders since both advanced age and an abnormal ORT may indicate reduced ovarian reserve and act as surrogate of ovarian stimulation cycle. in this case, the patients should be more properly defined as expected PORs

Exclusion Criteria:

* - Severe husband semen oligo terato atheno spermia
* Abnormal karyotyping of one or both couples
* Congenital and acquired uterine abnormalities
* Antiphospholipid Antibody syndrome
* Untreated hydrosalpinx
* Women intending to do PGD or screening
* Thin endometrium (< 7 mm) at day of HCG
* Premature luteinization (P> 2 ng/ml or P/E2 ratio > 1 on the day of HCG)
* Ovarian follicle > 10 mm and/or E2 > 40 pg/ml at day2 of stimulation cycle
* Less than two follicles (≥ 17mm) and/or E2 < 500 pg/ml at day of HCG

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 520 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
ongoing pregnancy rates | 20 weeks
  number of pregnancies completing 20 weeks or more gestational age expressed per patient

SECONDARY OUTCOMES:
clinical pregnancy rate | 8 weeks
  number of clinical pregnancies evidenced by ultrasound visualization of a gestational sac and embryonic pole with heart beat expressed per patient
miscarriage rate | 24 weeks
  number of pregnancies not completing 24 weeks of gestation

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - ART unit - Ain Shams university Matrnity Hospital, Cairo
  - Private fertility care centers, Cairo